CLINICAL TRIAL: NCT05330910
Title: A Randomized Controlled Trial Evaluating PAtients With Lax Gastroesophageal Junction to Initial Sleeve Gastrectomy With or Without Concomitant Crural Repair (REPAIR)
Brief Title: Crural Repair During Laparoscopic Sleeve Gastrectomy in Patients With a Lax Gastroesophageal Junction
Acronym: REPAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Chue Koy Min, Associate Consultant, Sengkang General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/2028
Record Dates: First submitted 2022-03-27; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Bariatric Surgery Candidate; Esophagus Injury; Gastroesophageal Reflux
Keywords: Obesity; Bariatric Surgery; Esophagitis; Gastroesophageal reflux disease; Laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux; Esophagitis

STUDY DESIGN:
Intervention Model Description: This study will be a double institution, double-blinded, randomized controlled trial, involving surgeons from the Upper Gastrointestinal and Bariatric Service, Department of General Surgery, Sengkang General Hospital (SKH) as well as the Department of Upper Gastrointestinal and Bariatric Surgery, Singapore General Hospital (SGH).
  Randomization will be performed by block randomization, with each block of 4. Block randomization was selected given the small study size, to ensure equal representation in both arms of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation concealment will be achieved via a central computer-generated random assignment, that will only be made known to the surgeon after the patient is induced on table prior to surgery. Participants from both institutions (SKH, SGH) will be within the same pool for block randomization, to ensure allocation concealment. Access or knowledge about the sequence of the randomization, will not be made known to the PI, Co-Is or mentor, and is only held by protocol administrator.
  Patient will be blinded to the randomization, and will only be told of the group of allocation at the end of completion of the study, at 1-year, after their postoperative endoscopy at 1-year. Outcomes assessor for primary outcomes at 1-year endoscopy will also be blinded to the initial surgery that was performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic sleeve gastrectomy arm (Active Comparator): Surgical technique will be standardized and will be performed by the study team. The bougie size for the LSG will be 40Fr, and a standard 5-port LSG will be performed. Standard protocolized postoperative recovery for all bariatric patients will be employed, including liquid diet with vitamins for the first 2 weeks postoperatively, followed by introduction of solid foods after.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy arm
- Laparoscopic sleeve gastrectomy with hiatal hernia repair arm (Experimental): Surgical technique will be standardized and will be performed by the study team. The bougie size for the LSG will be 40Fr, and a standard 5-port LSG will be performed. Standard protocolized postoperative recovery for all bariatric patients will be employed, including liquid diet with vitamins for the first 2 weeks postoperatively, followed by introduction of solid foods after. A hiatal dissection will also be performed during initial surgery, followed by a cruroplasty with Ethibon 0 sutures, in an interrupted manner.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy with concomitant hiatal hernia repair arm

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy with concomitant hiatal hernia repair arm — Surgical technique will be standardized and will be performed by the study team. The bougie size for the LSG will be 40Fr, and a standard 5-port LSG will be performed. Standard protocolized postoperative recovery for all bariatric patients will be employed, including liquid diet with vitamins for the first 2 weeks postoperatively, followed by introduction of solid foods after. A hiatal dissection will also be performed during initial surgery, followed by a cruroplasty with Ethibon 0 sutures, in an interrupted manner.
  Other Names: Laparoscopic sleeve gastrectomy with concomitant crural repair arm; Laparoscopic sleeve gastrectomy with concomitant cruroplasty arm
  Arms: Laparoscopic sleeve gastrectomy with hiatal hernia repair arm
Procedure: Laparoscopic sleeve gastrectomy arm — Surgical technique will be standardized and will be performed by the study team. The bougie size for the LSG will be 40Fr, and a standard 5-port LSG will be performed. Standard protocolized postoperative recovery for all bariatric patients will be employed, including liquid diet with vitamins for the first 2 weeks postoperatively, followed by introduction of solid foods after.
  Other Names: Laparoscopic sleeve gastrectomy; Laparoscopic sleeve gastrectomy alone
  Arms: Laparoscopic sleeve gastrectomy arm

SUMMARY:
Background:

Laparoscopic sleeve gastrectomy (LSG) is one of the commonest bariatric procedures. However, it is associated with postoperative gastroesophageal reflux disease (GERD) and erosive esophagitis (EE). The investigators' preliminary study suggests that the incidence of postoperative GERD and EE appears to be correlated with the preoperative presence of a lax gastroesophageal flap valve and hiatal hernia.

Hypothesis/ Aim:

To investigate the impact of a concomitant hiatal hernia repair with LSG on the incidence of postoperative EE.

Significance:

For patients with pre-existing EE, most surgeons will recommend a laparoscopic Roux-en-Y gastric bypass (LRYGB) as their primary bariatric procedure. However, compared to LSG, LRYGB is a technically more demanding procedure with increased morbidity and long term nutritional deficiencies. For asymptomatic patients at risk of postoperative EE due to presence of a hiatal hernia, there is still no consensus on the most appropriate bariatric surgical option. A LSG with a concomitant hiatal hernia repair, if shown to reduce EE postoperatively, may help to expand the pool of patients suitable for LSG in the future.

Methods:

A two center, double-blinded, randomized controlled trial of all patients, undergoing LSG with a preoperative diagnosis of a Hill's grade III gastroesophageal junction, will be randomized to having a concomitant hiatal hernia repair (experimental arm) versus just LSG alone (control arm). Primary outcome measures include 1-year postoperative EE on endoscopy. Secondary outcome measures include postoperative morbidity, blood loss, quality of life and GERD symptoms at 1-year postoperatively.

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy (LSG) is one of the most common bariatric procedures performed worldwide, accounting for more than 50% of all bariatric procedures, and with respectable weight loss and metabolic benefits which are comparable to the gold standard laparoscopic Roux-en-Y gastric bypass. However, one of the main disadvantages of LSG is its tendency to cause post-operative gastroesophageal reflux disease (GERD) and erosive esophagitis (EE).

To date, it is widely accepted that LSG should be avoided for patients with underlying GERD or EE. However, there is no consensus for asymptomatic patients, including those with an underlying hiatal hernia, which is known to predispose to GERD.

Currently, the two commonly employed methods for endoscopic classification of a hiatal hernia are via its axial length, or by grading the gastroesophageal flap valve, better known as the Hill's classification system.

Multiple retrospective cohort studies have documented a reduction in postoperative GERD following a concomitant LSG with a hiatal hernia repair, in patients with a preoperative diagnosed hiatal hernia. However, to date, there is only one randomized controlled trial which compared the efficacy of concomitant LSG with or without a concomitant hiatal hernia repair. Of the 100 patients, the trial did not report any differences in the incidence of postoperative GERD between the 2 groups. However, the trial had several limitations. Firstly, it included patients with no underlying hiatal hernia. In fact, of the 100 patients, 25 of them have no underlying hiatal hernia, thus may favour the outcome towards the null hypothesis. Subsequently, though the study attempted to randomize participants, while most baseline characteristics are well randomized, the most crucial element in the study, which was the length of the hiatal hernia, was significantly different between the 2 groups. Thirdly, the primary outcome was a subjective score via the Gastrointestinal Symptom Rating Scale (GSRS). Lastly, assessment of the presence of a hiatal hernia via the axial length is known to be operator-dependent, as well as subject to changes between inspiration and expiration, which can make its assessment less objective.

The investigators' propose using the alternative classification system for grading a hiatal hernia, called the Hill's classification system, to determine the preoperative hiatal laxity of the gastroesophageal flap valve, to determine which patients will likely benefit from a LSG with a concomitant hiatal hernia repair. The system, first introduced by Hill et al in 1996, was derived from an observational study of 13 cadavers to determine the presence of an anti-reflux valve and hiatal hernia. In the absence of a hiatal hernia, the angle of His, defined as the acute angulation along the greater curve of the stomach where the esophagus enters the stomach, creates a flap valve mechanism. This laxity of this flap valve varies and can be objectively graded based on the Hill's classification. This classification has been shown to be superior to the axial measurement of a hiatal hernia in the endoscopic assessment of the gastroesophageal junction and its association with GERD.

The Hill's classification system is much more objective. The grade III gastroesophageal junction is easily and objectively assessed, with little inter-observer variability, by the presence of a failure of closure of the endoscope around the hiatus. Unlike patients with Hill's grade IV gastroesophageal junction with a frank hiatal hernia, these patients with a grade III gastroesophageal junction mainly have a lax junction, with at most a physiological (<3cm) hiatal hernia on axial length.

Thus, this study proposes using the Hill's classification system to assess the efficacy of a concomitant crural repair with LSG in patients with a lax gastroesophageal flap valve. The investigators' hypothesize that a select group of patients with an underlying lax gastroesophageal junction may benefit from a concomitant crural repair with LSG. This group of patients, with grade III gastroesophageal junction, who have a lax hiatus and a small or physiological hiatal hernia, may potentially the only patient group that may benefit from a laparoscopic hiatal hernia or crural repair.

Study design:

This study will be a double institution, double-blinded, randomized controlled trial, involving surgeons from the Upper Gastrointestinal and Bariatric Service, Department of General Surgery, Sengkang General Hospital (SKH) as well as the Department of Upper Gastrointestinal and Bariatric Surgery, Singapore General Hospital (SGH).

Study population:

Eligible patients will come from patients visiting the bariatric surgery consultation clinic from both SKH and SGH. Patients that are deemed eligible for bariatric surgery will always undergo a routine esophagogastroduodenoscopy as part of standard preoperative evaluation. Patients found on esophagogastroduodenoscopy preoperatively to have a Hill's grade 3 gastroesophageal flap valve, with no evidence of EE will then be recruited.

Included patients should be patients aged between 21-65 years old, able to provide informed consent, with Hill's grade III gastroesophageal junction, that have opted to undergo LSG.

Excluded patients will include patients who are unable or unwilling to provide informed consent, with contraindications to LSG, who have opted not for LSG, who had previous upper gastrointestinal surgery, who have preoperative documented EE on endoscopy, who are graded Hill's grade I, II or IV gastroesophageal junction on retroflexion view of the endoscope with the stomach fully distended.

Randomization:

Patients will be blinded to their randomization allocation. Their allocation will only be made known should there be any adverse event, as per ethical guidelines, or after their end of 1-year follow-up.

Outcome measures:

Primary outcome measures will be presence of EE at the end of their 1-year follow-up after 1-year endoscopy. Secondary outcome measures will include any differences in SF-36 quality of life questionnaire, differences in their Gastrointestinal Symptom Rating Scale, as well as a Quality of Life in Reflux and Dyspepsia questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old
* Able to provide informed consent
* Hill's grade III gastroesophageal junction on preoperative endoscopy
* Opted to undergo laparoscopic sleeve gastrectomy as their bariatric procedure

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Contraindications to laparoscopic sleeve gastrectomy
* Opted not to undergo laparoscopic sleeve gastrectomy
* Had previous upper gastrointestinal surgery
* Had documented erosive esophagitis on preoperative endoscopy
* Had Hill's grade I, II or IV gastroesophageal junction on preoperative endoscopy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of post-operative erosive esophagitis | 1-year
  Presence or absence of erosive esophagitis on endoscopy
Degree of Post-operative erosive esophagitis | 1-year
  Grading of erosive esophagitis on endoscopy, noted as absent, or grade A, B, C or D (based on the Los Angeles classification)

SECONDARY OUTCOMES:
General Quality of Life Scores | 3-month, 6-month, 9-month, 1-year
  36-item Short Form Survey. It is a commonly employed questionnaire to assess overall quality of life. It comprises 36 short questions, which directly translates into a 0-100 scoring system. The higher the scores, the better the quality of life.
Gastroesophageal reflux disease symptoms | 3-month, 6-month, 9-month, 1-year
  Gastrointestinal Symptom Rating Scale. It is a questionnaire assessing 5 different symptom clusters of gastrointestinal symptoms, namely Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. Each domain has a 7-point graded scale, where 1 represents no symptoms and 7 represents very troublesome symptoms. Hence, the higher the scores in a particular domain, the more troublesome the symptoms. In assessing the endpoint of gastroesophageal reflux disease symptoms, the domain of reflux in the GSRS questionnaire will be evaluated.
Dysphagia symptoms | 3-month, 6-month, 9-month, 1-year
  Gastrointestinal Symptom Rating Scale. It is a questionnaire assessing 5 different symptom clusters of gastrointestinal symptoms, namely Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. Each domain has a 7-point graded scale, where 1 represents no symptoms and 7 represents very troublesome symptoms. Hence, the higher the scores in a particular domain, the more troublesome the symptoms. In assessing the endpoint of dysphagia symptoms as the secondary outcome, the domain of indigestion in the GSRS questionnaire will be evaluated.
Gastrointestinal reflux disease specific quality of life scores | 3-month, 6-month, 9-month, 1-year
  Quality of Life in Reflux and Dyspepsia questionnaire (QOLRAD). The QOLRAD (reflux version) is a 25-item questionnaire specifically focusing on gastroesophageal reflux symptoms. It can be scored based on frequencies, from none of the time to all of the time, for each question. The higher the frequency, the more prevalent the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Baldwin Po Man Yeung, MBChB, FRCS, Principal Investigator — Sengkang General Hospital; Jeremy Tian Hui Tan, MBBS, FRACS, Principal Investigator — Singapore General Hospital; Koy Min Chue, MBBS, FRCSEd, Principal Investigator — Sengkang General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Unless there is Institutional Ethics Board approval and patient consent

REFERENCES:
- [Background] Berger ER, Huffman KM, Fraker T, Petrick AT, Brethauer SA, Hall BL, Ko CY, Morton JM. Prevalence and Risk Factors for Bariatric Surgery Readmissions: Findings From 130,007 Admissions in the Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program. Ann Surg. 2018 Jan;267(1):122-131. doi: 10.1097/SLA.0000000000002079. PMID 27849660
- [Background] Peterli R, Wolnerhanssen BK, Peters T, Vetter D, Kroll D, Borbely Y, Schultes B, Beglinger C, Drewe J, Schiesser M, Nett P, Bueter M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss in Patients With Morbid Obesity: The SM-BOSS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):255-265. doi: 10.1001/jama.2017.20897. PMID 29340679
- [Background] Salminen P, Helmio M, Ovaska J, Juuti A, Leivonen M, Peromaa-Haavisto P, Hurme S, Soinio M, Nuutila P, Victorzon M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss at 5 Years Among Patients With Morbid Obesity: The SLEEVEPASS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):241-254. doi: 10.1001/jama.2017.20313. PMID 29340676
- [Background] Yeung KTD, Penney N, Ashrafian L, Darzi A, Ashrafian H. Does Sleeve Gastrectomy Expose the Distal Esophagus to Severe Reflux?: A Systematic Review and Meta-analysis. Ann Surg. 2020 Feb;271(2):257-265. doi: 10.1097/SLA.0000000000003275. PMID 30921053
- [Background] Assalia A, Gagner M, Nedelcu M, Ramos AC, Nocca D. Gastroesophageal Reflux and Laparoscopic Sleeve Gastrectomy: Results of the First International Consensus Conference. Obes Surg. 2020 Oct;30(10):3695-3705. doi: 10.1007/s11695-020-04749-0. Epub 2020 Jun 12. PMID 32533520
- [Background] Sgouros SN, Mpakos D, Rodias M, Vassiliades K, Karakoidas C, Andrikopoulos E, Stefanidis G, Mantides A. Prevalence and axial length of hiatus hernia in patients, with nonerosive reflux disease: a prospective study. J Clin Gastroenterol. 2007 Oct;41(9):814-8. doi: 10.1097/01.mcg.0000225678.99346.65. PMID 17881926
- [Background] Hansdotter I, Bjor O, Andreasson A, Agreus L, Hellstrom P, Forsberg A, Talley NJ, Vieth M, Wallner B. Hill classification is superior to the axial length of a hiatal hernia for assessment of the mechanical anti-reflux barrier at the gastroesophageal junction. Endosc Int Open. 2016 Mar;4(3):E311-7. doi: 10.1055/s-0042-101021. Epub 2016 Feb 10. PMID 27004249
- [Background] Hill LD, Kozarek RA, Kraemer SJ, Aye RW, Mercer CD, Low DE, Pope CE 2nd. The gastroesophageal flap valve: in vitro and in vivo observations. Gastrointest Endosc. 1996 Nov;44(5):541-7. doi: 10.1016/s0016-5107(96)70006-8. PMID 8934159
- [Background] Mahawar KK, Carr WR, Jennings N, Balupuri S, Small PK. Simultaneous sleeve gastrectomy and hiatus hernia repair: a systematic review. Obes Surg. 2015 Jan;25(1):159-66. doi: 10.1007/s11695-014-1470-0. PMID 25348434
- [Background] Snyder B, Wilson E, Wilson T, Mehta S, Bajwa K, Klein C. A randomized trial comparing reflux symptoms in sleeve gastrectomy patients with or without hiatal hernia repair. Surg Obes Relat Dis. 2016 Nov;12(9):1681-1688. doi: 10.1016/j.soard.2016.09.004. Epub 2016 Sep 14. PMID 27989522
- [Background] Holloway RH. The anti-reflux barrier and mechanisms of gastro-oesophageal reflux. Baillieres Best Pract Res Clin Gastroenterol. 2000 Oct;14(5):681-99. doi: 10.1053/bega.2000.0118. PMID 11003803
- [Background] Thor KB, Hill LD, Mercer DD, Kozarek RD. Reappraisal of the flap valve mechanism in the gastroesophageal junction. A study of a new valvuloplasty procedure in cadavers. Acta Chir Scand. 1987 Jan;153(1):25-8. PMID 3577567
- [Background] Navarini D, Madalosso CAS, Tognon AP, Fornari F, Barao FR, Gurski RR. Predictive Factors of Gastroesophageal Reflux Disease in Bariatric Surgery: a Controlled Trial Comparing Sleeve Gastrectomy with Gastric Bypass. Obes Surg. 2020 Apr;30(4):1360-1367. doi: 10.1007/s11695-019-04286-5. PMID 32030616
- [Derived] Chue KM, Toh BC, Ong LWL, Kariyawasam GM, Wong WK, Lim CH, Tan JTH, Yeung BPM. Rationale and Trial Protocol for a Double-Blinded Randomized Controlled Trial to assess the Impact of a Concomitant Crural Repair during Laparoscopic Sleeve Gastrectomy in Patients with a Lax Gastroesophageal Junction without Frank Hiatal Hernia (REPAIR trial protocol). Eur Surg Res. 2024 Feb 27. doi: 10.1159/000538043. Online ahead of print. PMID 38412840